CLINICAL TRIAL: NCT06641388
Title: A Phase I Study Evaluating the Single Subcutaneous Injection of Ebronucimab With Different Production Processes in Chinese Healthy Male Subjects
Brief Title: A Study Evaluating the Single Subcutaneous Injection of Ebronucimab in Chinese Healthy Male Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK102-102
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects (HS)
Keywords: phase I; healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ebronucimab 150mg (after the change) (Experimental): Ebronucimab 150mg Single subcutaneous injection into the abdomen.
  Interventions: Drug: Ebronucimab
- Ebronucimab 150mg (before the change) (Experimental): Ebronucimab 150mg Single subcutaneous injection into the abdomen.
  Interventions: Drug: Ebronucimab

INTERVENTIONS:
Drug: Ebronucimab — Ebronucimab subcutaneous injection
  Arms: Ebronucimab 150mg (after the change)
Drug: Ebronucimab — Ebronucimab subcutaneous injection
  Arms: Ebronucimab 150mg (before the change)

SUMMARY:
This is a phase I clinical study to evaluate the pharmacokinetics (PK) similarity of single dose subcutaneous injection of Ebronucimab with different production processes in Chinese healthy male subjects.

DETAILED DESCRIPTION:
This is a randomized, parallel controlled, phase I clinical study to evaluate the pharmacokinetics (PK) similarity of single dose subcutaneous injection of Ebronucimab with different production processes in Chinese healthy male subjects. This study consists of two parts: pre-trial part and formal-trial part, with a planned enrollment of approximately 180 healthy male participants from China.

ELIGIBILITY:
Key Inclusion Criteria:

* Weight: 60~80kg; Body mass index (BMI) ≥ 19 and ≤ 26 kg /m2 for healthy Chinese male subjects.
* Subjects fully understand the purpose, content, process, and potential adverse events of the trial, voluntarily participate in the trial, and sign an informed consent form before any trial procedure begins.
* Low density lipoprotein cholesterol (LDL-C) levels ≥ 1.8mmol/L and ≤ 4.9mmol/L during screening.
* Subjects are able to communicate well with the investigator and understand the requirements of the study.

Key Exclusion Criteria:

* 12 months prior use of PCSK9 inhibitors treatment.
* Allergic to the components of Ebronucimab and any monoclonal antibodies.
* History of important organ transplantation (such as heart, lung, liver, kidney, etc.).
* Abnormal vital signs during screening period and before randomization.
* Drug abuse prior to screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) | Baseline till last follow-up visit( up to day 43 or day 57)
  Assess the AUC of Ebronucimab
Maximum (peak) plasma concentration (Cmax) | Baseline till last follow-up visit( up to day 43 or day 57)
  Assess the Cmax of Ebronucimab
Incidence of adverse events(AE) | From the time of signing the informed consent form till last follow-up visit( up to day 43 or day 57)
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Free protein convertase of proprotein convertase subtilisin/kexin type 9 (PCSK-9) | Baseline till last follow-up visit( up to day 43)
  Concentration and percentage change from baseline of free protein convertase PCSK-9
Immunogenicity index | Day 1 and Day 57
  Number and percentage of subjects with detectable anti drug antibodies (ADA) and neutralizing antibodies (Nab) after treatment.
PCSK-9 concentration | Day 1 and Day 57
  Percentage change in PCSK-9 concentration compared to baseline
Serum Low-density lipoprotein Cholesterol (LDL-C) concentration | Day 1 and Day 57
  The change value and percentage of serum LDL-C concentration compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No